CLINICAL TRIAL: NCT01735630
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Efficacy and Safety Study of Oral ELND005 for Treatment of Agitation and Aggression in Patients With Moderate to Severe Alzheimer's Disease
Brief Title: Efficacy and Safety Study of ELND005 as a Treatment for Agitation and Aggression in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELND005-AG201; 2012-004299-20 (EudraCT Number)
Record Dates: First submitted 2012-11-25; First posted 2012-11-28 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease
Keywords: Agitation; Aggression; patients
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Aggression | interventions — scyllitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELND005 (Experimental): ELND005 film coated tablets, BID for 12 weeks
  Interventions: Drug: ELND005
- Placebo (Placebo Comparator): Matched placebo BID for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ELND005
  Other Names: Scyllo-inositol
  Arms: ELND005
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether ELND005 is effective in treating symptoms of agitation and aggression in patients with Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Probable AD according to the National Institute on Aging- Alzheimer's Association (NIA-AA) guidelines (McKhann et al 2011).
* MMSE score of 5 to 24 (inclusive) at the Screening Visit.
* Has clinically significant agitation/aggression defined as Neuropsychiatric Inventory (NPI)-agitation/aggression subscore of ≥4.
* No response or suboptimal response to standard nonpharmacological interventions.

Exclusion Criteria:

* The agitation/aggression is attributable to concomitant medications, environmental conditions, or active medical or psychiatric condition.
* Current diagnosis of major depressive disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Text Revision (DSM IV TR).
* Has persistent and distressing psychotic symptoms (delusion and/or hallucinations) that require psychiatric hospitalization.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (53):
  - TransitionTIL Investigational Site, Birmingham, Alabama
  - TransitionTIL Investigational Site, Phoenix, Arizona
  - TransitionTIL Investigational Site, Encino, California
  - TransitionTIL Investigational Site, Escondido, California
  - TransitionTIL Investigational Site, Fresno, California
  - TransitionTIL Investigational Site, Irvine, California
  - TransitionTIL Investigational Site, Long Beach, California
  - TransitionTIL Investigational Site, Los Alamitos, California
  - TransitionTIL Investigational Site, Los Angeles, California
  - TransitionTIL Investigational Site, Newport Beach, California
  - TransitionTIL Investigational Site, Santa Ana, California
  - TransitionTIL Investigational Site, Norwalk, Connecticut
  - TransitionTIL Investigational Site, Washington D.C., District of Columbia
  - TransitionTIL Investigational Site, Atlantis, Florida
  - TransitionTIL Investigational Site, Deerfield Beach, Florida
  - TransitionTIL Investigational Site, Delray Beach, Florida
  - TransitionTIL Investigational Site, Lake Worth, Florida
  - TransitionTIL Investigational Site, Miami, Florida
  - TransitionTIL Investigational Site, Oakland Park, Florida
  - TransitionTIL Investigational Site, Orlando, Florida
  - TransitionTIL Investigational Site, Ormond Beach, Florida
  - TransitionTIL Investigational Site, Port Charlotte, Florida
  - TransitionTIL Investigational Site, Sarasota, Florida
  - TransitionTIL Investigational Site, Sunrise, Florida
  - TransitionTIL Investigational Site, Columbus, Georgia
  - TransitionTIL Investigational Site, Savannah, Georgia
  - TransitionTIL Investigational Site, Springfield, Illinois
  - TransitionTIL Investigational Site, Bangor, Maine
  - TransitionTIL Investigational Site, Easton, Maryland
  - TransitionTIL Investigational Site, Winchester, Massachusetts
  - TransitionTIL Investigational Site, Ann Arbor, Michigan
  - TransitionTIL Investigational Site, Paw Paw, Michigan
  - TransitionTIL Investigational Site, Saint Paul, Minnesota
  - TransitionTIL Investigational Site, Hattiesburg, Mississippi
  - TransitionTIL Investigational Site, Stratford, New Jersey
  - TransitionTIL Investigational Site, Rochester, New York
  - TransitionTIL Investigational Site, Charlotte, North Carolina
  - TransitionTIL Investigational Site, Durham, North Carolina
  - TransitionTIL Investigational Site, Wilmington, North Carolina
  - TransitionTIL Investigational Site, Winston-Salem, North Carolina
  - TransitionTIL Investigational Site, Oklahoma City, Oklahoma
  - TransitionTIL Investigational Site, Portland, Oregon
  - TransitionTIL Investigational Site, Abington, Pennsylvania
  - TransitionTIL Investigational Site, Jenkintown, Pennsylvania
  - TransitionTIL Investigational Site, Norristown, Pennsylvania
  - TransitionTIL Investigational Site, Philadelphia, Pennsylvania
  - TransitionTIL Investigational Site, Pittsburgh, Pennsylvania
  - TransitionTIL Investigational Site, North Charleston, South Carolina
  - TransitionTIL Investigational Site, Port Royal, South Carolina
  - TransitionTIL Investigational Site, Nashville, Tennessee
  - TransitionTIL Investigational Site, DeSoto, Texas
  - TransitionTIL Investigational Site, Richmond, Virginia
  - TransitionTIL Investigational Site, Bellevue, Washington
- Canada (4):
  - TransitionTIL Investigational Site, Calgary, Alberta
  - TransitionTIL Investigational Site, Kelowna, British Columbia
  - TransitionTIL Investigational Site, Toronto, Ontario
  - TransitionTIL Investigational Site, Regina, Saskatchewan
- Spain (5):
  - TransitionTIL Investigational Site, Elche, Alicante
  - TransitionTIL Investigational Site, Getxo, Biscay
  - TransitionTIL Investigational Site, Barcelona
  - TransitionTIL Investigational Site, Burgos
  - TransitionTIL Investigational Site, Madrid
- United Kingdom (2):
  - TransitionTIL Investigational Site, Bath
  - TransitionTIL Investigational Site, Swindon

RESULTS

PARTICIPANT FLOW:
Groups:
- ELND005: ELND005 film coated tablets, BID for 12 weeks
  ELND005
- Placebo: Matched placebo BID for 12 weeks
  Placebo
Period: Overall Study
Arm/Group | ELND005 | Placebo
Started | 175 | 175
Completed | 157 | 157
Not Completed | 18 | 18
Not completed — Adverse Event | 8 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Sponsor Decision | 2 | 1
Not completed — Withdrawal by Subject | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELND005 | Placebo | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 20 | 33
  >=65 years | 162 | 155 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.2 (7.89) | 75.9 (8.51) | 76.0 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 100 | 195
  Male | 80 | 75 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 22 | 39
  White | 155 | 151 | 306
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 10 | 17
  United States | 153 | 152 | 305
  United Kingdom | 2 | 3 | 5
  Spain | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in NPI-C Combined Agitation and Aggression Subscores (NPI-C A+A).
Description: The NPI-C (de Medeiros et al 2010) is a validated and reliable behavioral measure that assesses psychopathology in dementia subjects. It evaluates 14 neuropsychiatric disturbances common in dementia.Higher scores on the NPI-C are associated with a greater clinical severity of symptoms. The NPI-C Agitation and Aggression score ranges from 0-63. The analysis of the NPI-C A+A score was performed on the mITT population.
Time Frame: Week 12
Population: mITT
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ELND005 | Placebo
Number analyzed (Participants) | 157 | 155
units on a scale | -4.3 (0.7) | -4.2 (0.7)

2. Secondary Outcome: Change From Baseline in Modified-ADCS-CGIC Agitation Scores
Description: The Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) is a widely used scale for the global assessment of change in AD trials.It is a 7-point Likert scale that ranges from marked improvement scored as 1 to marked worsening scored as 7, with no change scored as 4. The range is from 1 to 7. Higher scores indicate worsening agitation.
Time Frame: Week 12
Population: mITT population with available data for Modified-ADCS-CGIC Agitation Scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ELND005 | Placebo
Number analyzed (Participants) | 156 | 157
units on a scale | 3.6 (0.1) | 3.4 (0.1)

3. Secondary Outcome: Change From Baseline in NPI Total Scores
Description: The NPI (Cummings et al 1994) is a behavioral measure that assesses psychopathology in dementia subjects. It evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, nighttime behavior disturbances, and appetite and eating abnormalities. Higher scores on the NPI are associated with greater frequency and severity of symptoms. The scale range is 0-144.
Time Frame: Week 12
Population: mITT population with available data for NPI Total Scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ELND005 | Placebo
Number analyzed (Participants) | 157 | 154
units on a scale | -14.38 (1.69) | -15.12 (1.71)

4. Secondary Outcome: Change From Baseline in MMSE Scores
Description: The Mini-Mental State Exam (MMSE) (Folstein et al 1975) is a brief cognitive test assessing general cognitive function that has been employed in numerous clinical trials of products approved for the treatment of AD. The score can range from 0 to 30, with lower scores indicating greater impairment in function.
Time Frame: Week 12
Population: mITT population with available data for MMSE Scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ELND005 | Placebo
Number analyzed (Participants) | 157 | 154
units on a scale | -0.3 (0.2) | -0.4 (0.2)

5. Secondary Outcome: Change From Baseline in ADCS-ADL Scores
Description: The Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) (Galasko et al 1997) is a functional assessment that measures instrumental and basic activities of daily living. The total score for the 23-item ADCS-ADL ranges from 0 to 78 points, with lower scores indicating greater impairment in function.
Time Frame: Week 12
Population: mITT population with available data for ADCS-ADL Scores
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ELND005 | Placebo
Number analyzed (Participants) | 156 | 155
units on a scale | -1.458 (0.7) | -2.229 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient starting from the time the consent form was signed until the completion of the study
Arm/Group | ELND005 | Placebo
Serious Adverse Events (participants affected / at risk) | 17/175 | 5/175
Other Adverse Events (participants affected / at risk) | 97/175 | 82/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELND005 (N=175) | Placebo (N=175)
Fall (Injury, poisoning and procedural complications) | 2 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Homocidal ideation (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELND005 (N=175) | Placebo (N=175)
Agitation (Psychiatric disorders) | 14 | 13
Insomnia (Psychiatric disorders) | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 14 | 5
Vomiting (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 4 | 2
Urinary tract infection (Infections and infestations) | 12 | 7
Bronchitis (Infections and infestations) | 2 | 5
Dizziness (Nervous system disorders) | 2 | 7
Lethargy (Nervous system disorders) | 6 | 2
Somnolence (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 11 | 9
Contusion (Injury, poisoning and procedural complications) | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4
Gait disturbance (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days